CLINICAL TRIAL: NCT05104411
Title: Comprehensive Rehabilitation in Severely Ill Inpatients With COVID-19: A Cohort Study in a Tertiary Hospital
Brief Title: Rehabilitation in Severely Ill Inpatients With COVID-19
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Jaewon Beom, Clinical Associate Professor, Seoul National University Bundang Hospital
Other Study IDs: B-2108-705-112
Record Dates: First submitted 2021-10-22; First posted 2021-11-03 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: COVID-19
Keywords: Rehabilitation; Critical illness; Coronavirus disease 2019 (COVID-19_; Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2); Recovery of function
MeSH Terms: conditions — COVID-19; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Rehabilitative intervention — Active rehabilitation programs were done for all patients. Participants were asked to attend exercise program at PT room or bedside. Exercise program was offered once or twice daily on weekdays, by trained kinesiologists. In PT programs, most patients performed strengthening exercise of lower extremities, balance training, sit-up training, sit-to-stand training and gait training for about 30 minutes. Each program was individualized to participants' current physical function. In bedside programs, patients also underwent strengthening exercise and balance training without gait training for about 10 minutes. The duration of exercise program at PT room depends on the patient's condition(upto 1 month).

SUMMARY:
Inpatient rehabilitation of severe-to-critical COVID-19 patients(A longitudinal, single-center retrospective cohort)

DETAILED DESCRIPTION:
Patients who underwent intensive care at least two days and classified as severe-to-critical COVID-19 (WHO ordinal scale 5-7) were enrolled. Patients received comprehensive rehabilitation including active exercise program, nutritional support, and psychological support.

ELIGIBILITY:
Inclusion Criteria:

COVID-19 patients who

1. underwent intensive care at least two days,
2. eventually got negative conversion with two consecutive tests,
3. were classified as severe COVID-19 (WHO ordinal scale 5-7) and
4. participated in the inpatient rehabilitation program were included.

Exclusion Criteria:

COVID-19 patients who died (WHO ordinal scale 8) before discharge were excluded

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Severe COVID-19 (WHO ordinal scale 5-7) who participated in the inpatient rehabilitation program
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2021-08-14 (Actual); Primary Completion 2021-09-08 (Actual); Study Completion 2022-07-15 (Actual)

PRIMARY OUTCOMES:
Change of Functional Ambulation Classification | at baseline, immediately after rehabilitation completion, and 1-month after rehabilitation completion
  0~5 score. FAC 0(Nonfunctional ambulator), FAC1(Ambulator, dependent on physical assistance - Indicates a patient who requires continuous manual contact to support body weight as well as to maintain balance or to assist coordination), FAC 2(Ambulator, dependent on physical assistance - Indicates a patient who requires intermittent or continuous light touch to assist balance or coordination), FAC3(Ambulator, dependent on supervision), FAC4(Ambulator, independent level surface only), FAC5(Ambulator, independent). Higher score means better outcome.

SECONDARY OUTCOMES:
Change of Appendicular skeletal muscle mass index (ASMI) | at baseline, immediately after rehabilitation completion, and 1-month after rehabilitation completion
  [Kilogram Per Square Meter]
Change of Medical Research Council (MRC) sum score | at baseline, immediately after rehabilitation completion, and 1-month after rehabilitation completion
  0~60 score.
Change of handgrip strength | at baseline, immediately after rehabilitation completion, and 1-month after rehabilitation completion
  [Lb].
Change of number of 1-min sit-to-stand | at baseline, immediately after rehabilitation completion, and 1-month after rehabilitation completion
  Number of repetitions of sit-to-stand within one minute. Higher score means better outcome.
Change of walking speed | at baseline, immediately after rehabilitation completion, and 1-month after rehabilitation completion
  [meter per second]. Walking speed is measured by 10-meter walking test. If a patient cannot accomplish 10-meter walking test, 4-meter walking test is used instead. Higher score means better outcome.
Change of Berg balance scale | at baseline, immediately after rehabilitation completion, and 1-month after rehabilitation completion
  0~56 score. Berg balance scale is 14-item objective measure that assesses static balance and fall risk in adults. Each item consists of a five-point ordinal scale(0 to 4), with 0 indicating the lowest level of function and 4 the highest level of function. Higher score means better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jaewon Beom, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Woo H, Lee S, Lee HS, Chae HJ, Jung J, Song MJ, Lim SY, Lee YJ, Cho YJ, Kim ES, Kim HB, Lim JY, Song KH, Beom J. Comprehensive Rehabilitation in Severely Ill Inpatients With COVID-19: A Cohort Study in a Tertiary Hospital. J Korean Med Sci. 2022 Aug 29;37(34):e262. doi: 10.3346/jkms.2022.37.e262. PMID 36038958